CLINICAL TRIAL: NCT07141212
Title: Effect Of Virtual Reality On Pulmonary Function And Anxiety Levels In Asthmatic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mai Gomaa Mohamed Abdelrahman, Principal Investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Virtual Reality in Asthma
Record Dates: First submitted 2025-07-22; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko breathing exercise group (Active Comparator): The participant will participate in Buteyko breathing only twice\ week for 8 weeks and the session was about 10 min, with their optimal medical treatment,which depending on three steps:
  Step 1: The ''Control pause (CP)'' breathing test Step 2: Shallow breathing Sit up straight Step 3: Putting it together Take Control pause
  Interventions: Procedure: Buteyko Breathing
- Virtual Reality group (Experimental): The participants will receive 20 min VR and Buteyko breathing along with prescribed medical treatment for 8 weeks , twice \week. Training depends on two breathing training aspects with 5 breathing cycles for each one, 30 sec rest in between. in form of: Colour Breathing VR program (Box Breathing), LAMINAL VR (Calm).
  Interventions: Device: Virtual reality glass

INTERVENTIONS:
Device: Virtual reality glass — Virtual reality (VR), with its immersion and interactivity, offers the possibility to amplify the effectiveness of breathing techniques in promoting mental health by creation of relaxing scenarios and has been successfully employed in promoting relaxation and stress reduction. Virtual reality can turn breathing exercises into an interactive experience that feels more like a fun activity than a tedious task. It consists of VR headset, two touch controllers, glasses spacer with adjustable straps for good vision as follows:
  1. Colour Breathing VR program (Box Breathing) :
     Patient sit in comfortable position with relaxed both shoulders. Breath in for 4 second, Hold breath for 4 sec, Breath out for 4 sec, Hold for 4 sec, Inhalations and exhalations move a 3D cloud shaped object closer and farther away from the user.
  2. LAMINAL VR (Calm): Inhalations and exhalations grow and shrink a 2D circle with bubbles in between, changing in color.
  Arms: Virtual Reality group
Procedure: Buteyko Breathing — 1. The ''Control pause (CP)'' breathing test: Hold his nose on the "out" breath, with empty lungs but not too empty and count how many seconds that he can comfortably last before the need to breathe in again.
  2. Shallow breathing Sit up straight: breathe air slightly into the tip of the nostrils. Concentrate on calming his breath to reduce the amount of warm air he feel on his finger, try to maintain the need for air for about 4 min.
  3. Putting it together Take Control pause:
  Reduced breathing for 4 min. Wait 2 min and take Control pause. Reduced breathing for 4 min. Wait 2 min and take Control pause.
  Arms: Buteyko breathing exercise group

SUMMARY:
The Purpose of the Study This study will be conducted to determine the effect of virtual reality on pulmonary function and anxiety levels in moderate to severe asthmatic patients.

DETAILED DESCRIPTION:
Globally, asthma is the 16th cause of years-lived with-disability and the 28th most common source of burden of disease; it accounts for 1 in every 250 deaths. In Egypt, over 6.7% and 26.5% of the general adult and pediatric population, respectively, have asthma. At least 1/3 of the patients with persistent asthma experience symptoms of anxiety/depression. There is a lack of data regarding other asthma subgroups, namely adolescents and those with mild or moderate persistent asthma.

Recently, there has been a global concern for the treatment of asthma through physical therapy and complementary alternative medicine (CAM). Buteyko breathing technique is one of CAM techniques that is becoming more prevalent.

Virtual reality is an emerging new technology that has drawn scientists' attention to its potential impact on rehabilitation. It is a safe and effective medium for supporting stress and anxiety management.

In general, the literature has shown that VR This would enable users to learn over time how to change their physiological activity to enhance health and performance, reduce stress-related symptoms, and increase their well-being.

Up to investigated knowledge, No previous studies conducted to explore the effect of VR on pulmonary function and anxiety in adult patients with moderate to sever bronchial asthma.

HYPOTHESES: It will be hypothesized that there will be no significant effect of Virtual Reality on pulmonary function and anxiety levels in patients with moderate to sever bronchial asthma.

RESERCH QUESTION: Does virtual reality affect pulmonary function and anxiety levels in moderate to severe asthmatic patients?

ELIGIBILITY:
Inclusion Criteria:

* Both sexes would be previously diagnosed as bronchial asthma with a cut-off score FEV1: Between 60% and 80% of predicted value or less than 60% of predicted value and FEV1/FVC ratio: May be significantly reduced from normal value 0.75-0.80.
* The age of the patients will be ranged between 30 and 40 years old.
* Asthma Control Test(ACT) will be less than 16 can be successfully used to identify those who will be uncontrolled asthma.
* All patients will be assessed by Hospital Anxiety and Depression Scale (HADS) ;A cut-off score of 11-15 a moderate depression/anxiety level.
* Patients who are conscious and cooperative.
* Patients who are able to understand and follow instruction.

Exclusion Criteria:

* Previous participation in any pulmonary rehabilitation program.
* Cardiovascular instabilities such as: Uncontrolled hypertension, Uncontrolled arrhythmia and Recent ischemic event.
* Mental disorders preventing protocol implementation.
* Other chronic respiratory diseases.
* Pregnant women.
* New or current smoker.
* Respiratory tract infection.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Control pause breathing test | 8 weeks
  It is part of the Buteyko method of breathing exercises and is designed to measure the length of time a person can comfortably hold their breath after a normal exhalation. its normal range is between 0-60 seconds, less than 20 seconds means poor control.
Asthma control test | 8 weeks
  It was a commonly valuable tool to assess asthma control that typically involves a self-reported questionnaire that evaluates symptoms over the past 4 weeks. It is self reported 5-25 scale. Higher score indicates better control. less than 16 indicates uncolntrolled asthma
Forced Expiratory Volume in one second (FEV1) | 8 weeks
  FEV1 stands for Forced Expiratory Volume in 1 second. It is a measurement taken during a spirometry test, which assesses lung function. Specifically, it measures the amount of air a person can forcefully exhale in the first second of a forced exhalation. A lower FEV1 reading can indicate an obstruction in the airways, potentially pointing to conditions like asthma. Normal values for % predicted FEV1 are generally 80% or higher of the predicted value. 60-80%moderate, <60% severe.
Forced vital capacity (FVC) | 8 weeks
  Forced vital capacity (FVC) is the maximum amount of air a person can exhale after taking the deepest possible breath. It's a key measurement in spirometry, a common breathing test used to assess lung function. FVC helps doctors identify and distinguish between different types of lung diseases, including obstructive (like asthma). FVC can also be expressed as a percentage of the predicted value, with 80% to 120% considered within the normal range
FEV1/FVC ratio | 8 weeks
  The FEV1/FVC ratio is a calculation used in pulmonary function tests, specifically spirometry, to assess lung function. It represents the proportion of a person's forced vital capacity (FVC) that they can exhale in the first second of a forced expiration, known as forced expiratory volume in 1 second (FEV1). A normal FEV1/FVC ratio is typically above 70% (0.75-0.80), and a lower ratio suggests an airway obstruction
Peak expiratory flow (% predicted) | 8 weeks
  It refers to the percentage of a person's measured PEF compared to their predicted PEF, based on factors like age, sex, and height. It's a way to assess how well someone is breathing compared to what's expected for them, with lower percentages often indicating airflow obstruction such as asthma. PEF predicted % is calculated by dividing the actual PEF measurement by the predicted PEF and multiplying by 100.
  A lower PEF predicted % generally indicates a greater degree of airflow obstruction.
  For example, in asthma, a PEF predicted % below 50% may indicate a severe exacerbation.
Anxiety level by Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  It is a 14-item questionnaire that assesses anxiety and depression symptoms for all participants before and after the treatment program. It has two seven-item subscales, one for anxiety and one for depression. Each item is scored on a 4-point scale, with a maximum score of 21 for each subscale. Scores are categorized as normal (0-7), mild (8-10), moderate (11-14), and severe (15-21) for both anxiety and depression.

SECONDARY OUTCOMES:
Treatment Adherence Perception Questionnaire(TAPQ) | 8 weeks
  It is a new, brief self-report instrument for assessing patient perceptions and attitudes regarding their own adherence to medical treatment plans. It consists of three distinct scales: Perceived Behavior, Perceived Benefit, and Perceived Burden. Each scale is scored using a Likert-type scale, and higher scores generally indicate more positive perceptions of adherence. Each scale typically contains a set number of items (e.g., 5 items). These items are rated on a Likert-type scale, such as:1 = Strongly Disagree, 2 = Disagree, 3 = Uncertain, 4 = Agree, 5 = Strongly Agree. The scores for each item within a scale are summed to produce a total score for that scale.
Functional capacity | 8 weeks
  It is measured by the 6-minute walk test; it is a simple, standardized assessment of functional exercise capacity, particularly useful for individuals with cardiopulmonary conditions. It measures the distance a patient can walk in six minutes, providing insights into their overall exercise tolerance and response to exertion. Less than 3 minutes walking or associated symptoms like fatigue, pain, or dyspnea indicate reduced functional capacity.
Frequency of exacerbations (time/day) | 8 weeks
  It can refer to how often asthma exacerbation occurs within a single day. exacerbations are defined as worsening symptoms of breathlessness, cough, and/or sputum production, and they can be triggered by various factors like infections or air pollution. Frequent exacerbations are a hallmark of severe asthma and can significantly impact a patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra M Serry, As Professor, Study Chair — Cairo University; Donia M El Masry, Lecturer, Study Director — Cairo University; Karim A Fathy, Professor, Principal Investigator — Faculty of Physical therapy October 6 University; Amira I Alam Eldin, As Professor, Principal Investigator — Cairo University
Locations (1):
- October 6 university hospital outpatient chest department, Giza, Cairo Governorate, Egypt

REFERENCES:
- [Background] Esposito C, Autorino G, Iervolino A, Vozzella EA, Cerulo M, Esposito G, Coppola V, Carulli R, Cortese G, Gallo L, Escolino M. Efficacy of a Virtual Reality Program in Pediatric Surgery to Reduce Anxiety and Distress Symptoms in the Preoperative Phase: A Prospective Randomized Clinical Trial. J Laparoendosc Adv Surg Tech A. 2022 Feb;32(2):197-203. doi: 10.1089/lap.2021.0566. Epub 2021 Dec 28. PMID 34962159